CLINICAL TRIAL: NCT05236621
Title: A Multicenter, Open-Label, Single-Arm Clinical Study of the Efficacy and Safety of Pomalidomide Capsules Combined With Low-Dose Dexamethasone in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of the Efficacy and Safety of Pomalidomide Capsules Combined With Low-Dose Dexamethasone in Subjects With Relapsed and Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-YK4-056-003
Record Dates: First submitted 2022-01-24; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma; Recurrent or Refractory
Keywords: Permadomide capsules
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Permadomide + Low-Dose Dexamethasone (Experimental): Participants received 4 mg pomalidomide administered by mouth on Days 1 to 21 of each 28-day treatment cycle and 40 mg dexamethasone administered by mouth once per day on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — 4 mg pomalidomide capsules administered orally
Drug: Dexamethasone — 40 mg dexamethasone tablets administered orally

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of permadomide capsules developed by Qilu Pharmaceutical Co., LTD.

ELIGIBILITY:
Inclusion Criteria:

1.Subjects diagnosed with multiple myeloma according to the diagnostic criteria of Chinese Multiple Myeloma Diagnosis and Treatment Guidelines (Revised in 2020); 2.Must be ≥ 18 years of age,male or female, if the subject is of childbearing age and should use effective contraceptive methods, the subject must agree to comply with all contraceptive requirements:

1. there are fertile women have to decide, at the same time take two reliable contraceptive methods (an effective contraceptive method is: tubal ligation, intrauterine contraceptive device, hormone (birth control pills, needles, patch, vaginal ring or implants) or partner vasectomy, another effective birth control method is: male or synthetic rubber condom, diaphragm or cervical cap). Unless hysterectomy is performed, effective contraception is required even if there is a history of infertility.
2. Fertile men must use rubber or synthetic condoms at all times during the use of this product and during sexual contact with fertile women within 28 days of discontinuation of this product, even if participants have successfully had a vasectomy.

3. Received at least two previous treatments (in different treatment regimens or the same regimen, including at least 2 cycles of lenalidomide and 2 cycles of proteasome inhibitors [such as bortezomib or ixazomib]) Relapse of multiple myeloma or ineffective to the last treatment (definition of last treatment ineffective: disease progression during the use of the treatment plan or disease progression within 60 days after the completion of the treatment plan), the last treatment plan is not limited; 4. Multiple myeloma subjects with measurable M protein, i.e., at least one of the following 3 assays:

1. Serum M protein≥0.5g/dL (5g/L);
2. Urine M protein≥200mg/24h;
3. Determination of serum free light chain: in the case of abnormal serum free light chain ratio, the level of involved free light chain is ≥10 mg/dL (100 mg/L); 5. Hematology meets the following conditions:

1) ANC≥1.0 x10^9/L (including ANC≥1.0x10^9/L supported by G-CSF); 2) PLT≥50 x10^9/L； 3) When plasma cells in bone marrow ≥50%, no specific requirements for neutrophil count, platelet ≥30 x10^9/L can be selected; 6. Liver and kidney function tests meet the following conditions:

1. TBIL ≤ 2.0mg/dL；
2. ALT、AST ≤ 3.0 x ULN； 3) Serum creatinine ≤ 3.0 mg/dL or creatinine clearance rate ≥ 30 mL/min; 7. Those who can accept and can use antithrombotic drugs, such as low molecular weight heparin sodium or aspirin; 8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2, expected survival ≥ 3 months; 9. There must be a washout period of ≥ 2 weeks (14 days) from the last treatment (excluding dexamethasone treatment); 10. Subjects voluntarily joined the study and signed a written informed consent.

Exclusion Criteria:

1. Subjects who cannot tolerate thalidomide, lenalidomide, pomalidomide and other types of drug treatment according to the judgment of the investigator.
2. Subjects who have had allergic reactions to immunomodulators similar to pomalidomide, dexamethasone or components contained in the drug;
3. Diagnosis of non-secretory MM (non-secretory subjects or subjects with a small amount of free light chain but less than 100mg/L) in multiple myeloma;
4. Subjects with active new thrombosis or unwilling to undergo antithrombotic therapy;
5. The subjects are suffering from other tumors at the same time or have a past history of tumors, or have undergone anti-tumor treatment (including major surgery) within the last 4 weeks, except for the following tumor diseases or those who have lived without tumors for ≥ 3 years so far: skin base Cell carcinoma, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histologic findings of prostate cancer (TNM clinical stage T1a or T1b), or treated prostate cancer;
6. Subjects suffering from central nervous system diseases and requiring treatment;
7. Subjects with peripheral neuropathy ≥ grade 3;
8. Subjects who need to use immunosuppressive or steroid drugs for a long time;
9. Known subjects with hepatitis B virus (HBV-DNA ≥ 1×10^3 copies/mL or HBV-DNA > 200 IU/mL) or hepatitis C virus (HCV) activity, or human immunodeficiency virus (HIV) ) serologically positive;
10. Subject has any of the following:

1) According to the NYHA classification standard, cardiac insufficiency grade 2 or above; 2) Myocardial infarction occurred within one year; 3) poorly controlled angina pectoris, including variant angina pectoris; 11. Subjects have serious infectious diseases at the same time; 12. Subjects planning to become pregnant or unable to take reliable contraceptive measures; 13. Women who are pregnant or breastfeeding; 14. Subjects who have received allogeneic hematopoietic stem cell transplantation within 12 months, or who have active graft-versus-host disease (GVHD) or who require immunosuppressive therapy after 12 months of allogeneic hematopoietic stem cell transplantation； 15. Those who participated in other clinical trials and received experimental drugs within one month before the first drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Total Response Rate(ORR) | From randomization through the study follow-up phase; up to the data cut-off of 1 December 2023; Maximum time on follow-up was 104 weeks.
  Statistical analysis of ORR of primary efficacy will be based on IRC remission assessment results, as well as the investigator's remission assessment.Strict Complete Response (sCR) + Complete Response (CR) + Partial Response (PR) + Very Good PR (VGPR).

SECONDARY OUTCOMES:
Duration of remission(DoR) | The time from the first observation of at least partial remission (PR) to disease progression (PD) or death from any cause is whichever comes first, assessed up to 104 weeks.
  The time from the first observation of at least partial remission (PR) to disease progression (PD) or death from any cause is whichever comes first.
Progression-free survival(PFS) | up to 104 weeks
  The time between the first dose of this trial and the onset of progression (evaluated according to IMWG efficacy criteria listed in the China Guidelines for the Diagnosis and Treatment of Multiple Myeloma 2020 (see attachment)) or death.
Overall survival(OS) | up to 104 weeks
  The time between enrollment for the first dose of the study and the death of the patient from any cause (the last follow-up date for the lost subjects and the end date for the patients who were still alive at the end of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Chen, MD, PhD, Principal Investigator — Beijing Chao Yang Hospital; Juan Li, MD, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Hongmei Jing, MD, PhD, Principal Investigator — Peking University Third Hospital; Huo Tan, MD, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Shunqing Wang, MD, PhD, Principal Investigator — Guangzhou First People's Hospital; Ying Zhao, MD, PhD, Principal Investigator — First People's Hospital of Foshan; Xun Lai, MD, PhD, Principal Investigator — Yunnan Cancer Hospital; Qing Wang, MD, PhD, Principal Investigator — Guizhou Provincial People's Hospital; Jinqiao Zhang, MD, PhD, Principal Investigator — Hebei Medical University Third Hospital; Lihong Liu, MD, PhD, Principal Investigator — Hebei Medical University Fourth Hospital; Baijun Fang, MD, PhD, Principal Investigator — Henan Tumor Hospital; Junjun Li, MD, PhD, Principal Investigator — The First Affiliated Hospital of Nanhua University; Binghua Wang, MD, PhD, Principal Investigator — Weihai Central Hospital; Wei Yang, MD, PhD, Principal Investigator — Shengjing Hospital; Wei Wang, MD, PhD, Principal Investigator — The Affiliated Hospital of Qingdao University; Ming Hou, MD, PhD, Principal Investigator — Shandong University Qilu Hospital; Aili He, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi 'an Jiaotong University; Yafei Wang, MD, PhD, Principal Investigator — Tianjin Cancer Hospital; Jie Jin, MD, PhD, Principal Investigator — The First Affiliated Hospital of Zhejiang University Medical College (Hematology); Xuehong Ran, MD, PhD, Principal Investigator — Weifang People's Hospital; Jiao Chen, MD, PhD, Principal Investigator — Sichuan Provincial People's Hospital; Liping Su, MD, PhD, Principal Investigator — Shanxi Province Cancer Hospital; Yanping Ma, MD, PhD, Principal Investigator — Second Hospital of Shanxi Medical University; Yanping Song, MD, PhD, Principal Investigator — Xi 'an Central Hospital; Congmeng Lin, MD, PhD, Principal Investigator — Zhangzhou Hospital, Fujian Province; Quanyi Lu, MD, PhD, Principal Investigator — Zhongshan Hospital Xiamen University; Da Gao, MD, PhD, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Wenhong Lai, MD, PhD, Principal Investigator — The First Affiliated Hospital of Gannan Medical College; Jianping Hao, MD, PhD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Taiwu Xiao, MD, PhD, Principal Investigator — Liaocheng People's Hospital; Zhen Cai, MD, PhD, Principal Investigator — The First Affiliated Hospital of Zhejiang University Medical College (Transplant Center); Xin Zhou, MD, PhD, Principal Investigator — Wuxi People's Hospital
Locations (23):
- China (23):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Shengjing Hospital affiliated to China Medical University, Beijing, Beijing Municipality
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Tumor Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Second Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University Medical College (Hematology), Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhou H, Wang Y, Chen J, He A, Jin J, Lu Q, Zhao Y, Li J, Hou M, Su L, Lai X, Wang W, Liu L, Ma Y, Gao D, Lai W, Zhou X, Jing H, Zhang J, Yang W, Ran X, Lin C, Hao J, Xiao T, Huang Z, Zhu Z, Wang Q, Fang B, Wang B, Song Y, Cai Z, Liu B, Zhu Y, Yang X, Kang X, Li J, Chen W. Efficacy and safety of generic pomalidomide plus low-dose dexamethasone in relapsed or refractory multiple myeloma: a multicenter, open-label, single-arm trial. Ann Hematol. 2024 Mar;103(3):855-868. doi: 10.1007/s00277-023-05558-y. Epub 2023 Dec 19. PMID 38112795